CLINICAL TRIAL: NCT06806098
Title: Cessation Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Responsible Party: Principal Investigator, Amanda L. Graham, PhD, Chief Health Officer, Truth Initiative
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CessationClinicalTrial
Record Dates: First submitted 2024-11-13; First posted 2025-02-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Use Cessation
Keywords: Digital intervention
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Data collection staff will be blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sponsored cessation intervention (Experimental): Intervention arm receiving sponsored version only available for enterprise client users.
  Interventions: Behavioral: Truth Initiative Digital Cessation Program
- Usual Care (Active Comparator): Usual care control arm receiving referral to a free digital cessation program
  Interventions: Behavioral: Usual Care
- Free cessation intervention (Experimental): Intervention arm receiving free version of a cessation intervention.
  Interventions: Behavioral: Truth Initiative Digital Cessation Program
- Assessment-only (No Intervention): Periodic assessment check-ins only, no active intervention

INTERVENTIONS:
Behavioral: Truth Initiative Digital Cessation Program — Truth Initiative's digital cessation program is a multimodal evidence-based, digital tobacco cessation program. Accessible on any web-enabled device, it was developed with the Mayo Clinic around tobacco dependence treatment guidelines, Social Cognitive Theory, and the Mayo Clinic model for engaging tobacco users in cessation treatment. It includes a personalized quit plan with AI-driven content recommendations, interactive exercises, educational videos, and emails; a dynamically tailored, bidirectional text message program; the longest-running online community dedicated to tobacco cessation; synchronous live chat coaching (sponsored version only); and pharmacotherapy decision support and delivery (sponsored version only).
  Arms: Free cessation intervention; Sponsored cessation intervention
Behavioral: Usual Care — Smokefree.gov is a web-based tobacco cessation platform run by the National Cancer Institute of the National Institutes of Health since 2003 and represents the current standard of care for digital tobacco cessation in the U.S. As of 2020, the SmokeFree.gov Initiative (SFGI) consisted of a multimodal suite of interventions - 6 mobile-optimized websites, 9 text messaging programs, 2 mobile apps, and social media platforms.
  Arms: Usual Care

SUMMARY:
The Cessation Clinical Trial will investigate the effectiveness of a digital quit tobacco program in promoting abstinence from tobacco product use compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Current tobacco use (past 30-day use of one or more of the following: cigarettes, cigars, little cigars, cigarillos, e-cigarettes, or oral nicotine products)
* US residence
* Active text message plan (phase 2 only)

Exclusion Criteria:

* Age 25 or above (phase 2 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2220 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
30-day point prevalent abstinence | 7-months post randomization
  30-day point prevalent abstinence from user's primary product to quit indicated at enrollment

SECONDARY OUTCOMES:
Abstinence from all tobacco products | 7 months post randomization
  Abstinence from any combustible tobacco product and any nicotine-containing product.
  Past 30-day abstinence will be measured for the following tobacco/nicotine products one by one and a combined total abstinence measure will be calculated based on these responses.
  Measurement item:
  In the past 30 days, which of the following products have you used at all (i.e., even a puff/hit)? Response options are Yes/No for each item.
  * Cigarettes
  * E-cigarettes
  * Chew
  * Dip
  * Nicotine pouches
  * Cigars/little cigars/cigarillos

CONTACTS AND LOCATIONS:
Locations (1):
- Truth Initiative, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified dataset will be available for replication purposes with a Data Sharing Agreement with Truth Initiative.